CLINICAL TRIAL: NCT01287182
Title: Trial of Ateronon in Patients With Coronary Disease to Evaluate Its Effectiveness in Assessing the Risk Factors of Atherosclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omicron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP2912011
Record Dates: First submitted 2011-01-29; First posted 2011-02-01 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Atherosclerosis
Keywords: Asymptomatic Myocardial Ischemic patients
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
- Ateronon (Active Comparator)
  Interventions: Drug: Ateronon

INTERVENTIONS:
Drug: Ateronon — Ateronon daily for 3 months
  Arms: Ateronon

SUMMARY:
This is a trial of Ateronon in Patients with Coronary Disease to Evaluate its Effectiveness in Assessing the Risk Factors of Atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women with demonstrated Coronary Disease
* AtheroAbzyme positive during screening process
* Elevated Total Cholesterol
* Willingness to take study nutritional supplement once a day for 3 months

Exclusion Criteria:

* Women who are pregnant, nursing or intend pregnancy during the period of treatment
* Known milk, soy or whey allergy

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
to evaluate the effectiveness of Ateronon in inhibiting atherogenic lipid oxidation in patients with demonstrated coronary disease | Baseline and 3 months

SECONDARY OUTCOMES:
to evaluate the potential effectiveness of Ateronon in lowering pulse rate as well systolic and diastolic blood pressure in patients with demonstrated coronary disease | Baseline and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rafic Hariri University Hospital, Beirut, Bir Hasan, Lebanon